CLINICAL TRIAL: NCT02143284
Title: Single-Center, Exploratory Study of EndoChoice's Upper&Lower Endoscopic Systems Utilizing EndoChoice's Full Spectrum Optical Technology
Brief Title: A Study of EndoChoice's Upper&Lower Endoscopic Systems Utilizing a Full Spectrum Optical Technology
Acronym: FUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EndoChoice Innovation Center, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CD-1715
Record Dates: First submitted 2014-05-05; First posted 2014-05-21 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endoscopy exploratory single arm (Experimental): Exploratory single arm, the system will be used in otherwise standard procedures, and will be reviewed in terms of performance, usability, ease of use and safety.
  Interventions: Device: Endoscopy exploratory single arm (EndoChoice FUSE(TM) System)

INTERVENTIONS:
Device: Endoscopy exploratory single arm (EndoChoice FUSE(TM) System) — The investigational device will be applied in otherwise standard procedures (upper and lower Gastrointestinal tract endoscopy)

SUMMARY:
EndoChoice's FUSE System enables a wider view range via 1-2 additional cameras (depending on the model). These optical properties are to be examined and reviewed in this trial (mainly usability and safety)

DETAILED DESCRIPTION:
EndoChoice Full Spectrum Optical Technology (FSOT) in gastrointestinal endoscopy enables a 330 degree field of view. FSOT powers EndoChoice's FDA, CE and AMAR (Israeli medical device authority) approved Endoscopic systems (Gastroscope and Colonoscope). The intent of this study is to evaluate the safety, performance and usability of additional versions of FSOT- powered gastroscopes and colonoscopes.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients ages of 18-70
* The patient has been scheduled for routine screening upper or lower endoscopy, diagnostic endoscopic work up, or endoscopic surveillance.
* Signed informed consent

Exclusion Criteria:

* Patients with inflammatory bowel disease;
* Patients with a personal history of polyposis syndrome;
* Patients with suspected bowel stricture potentially precluding complete endoscopy
* Patients with a history of diverticulitis or toxic megacolon
* Patients with a history of radiation therapy to neck, abdomen, pelvis;
* Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.
* Patients with GI bleeding, that has not been corrected prior to endoscopy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Performance, usability and ease of use | 1 Year
  The performance of the device is assessed via a performance questionnaire which the recruiting (and treatment providing) physician will answer.

SECONDARY OUTCOMES:
Safety | 1 Year
  The safety of the device will be assessed as a secondary outcome measure according to quantity and nature of adverse and severe adverse events, if such occur.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Gralnek, Prof., Principal Investigator — Rambam Medical Center Gastroenterological institute
Locations (1):
- Rambam medical center, Haifa, Israel, Israel